CLINICAL TRIAL: NCT06357312
Title: Influence of Static Distal Locking on Outcomes of Unstable Intertrochanteric Fracture Treated With a Short Proximal Femoral Nail
Brief Title: Influence of Static Distal Locking of a Short Proximal Femoral Nail
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elda University Hospital (Other)
Responsible Party: Principal Investigator, Francisco Antonio Miralles-Muñoz, Head of Department of Orthopedic Surgery, Elda University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/11P
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Hip Fracture
Keywords: hip; fracture; intertrochanteric; elderly; screw
MeSH Terms: conditions — Hip Fractures; Fractures, Bone

STUDY DESIGN:
Intervention Model Description: Prospective, comparative, randomized and double-blind study
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding of the patient included in the study and the investigator evaluating the results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group with distal screw (Experimental): Patients who have been randomly selected for this procedure are included.
  Interventions: Device: hip trochanteric nail
- Group without distal screw (Experimental): Patients who have been randomly selected for this procedure are included.
  Interventions: Device: hip trochanteric nail

INTERVENTIONS:
Device: hip trochanteric nail — hip trochanteric nail with and without distal interlocking screw

SUMMARY:
Prospective, comparative, randomized, double-blind study to evaluate the outcomes of trochanteric nailing in unstable hip fractures with and without a distal interlocking screw.

DETAILED DESCRIPTION:
Due to the lack of first-level evidence, this study aims to evaluate the effectiveness and safety of surgical treatment for unstable hip fractures, with or without the inclusion of a distal interlocking screw in the hip nail.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 50 years old
* With unstable intertrochanteric hip fracture
* Operated in the first 48 hours after hospital admission

Exclusion Criteria:

* Simultaneous associated fractures
* Fractures with subtrochanteric line
* Non-acute fractures

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of functional status using the Barthel index | 12 months
  Evaluation of functional status 12 months after hip surgery

SECONDARY OUTCOMES:
Postoperative mechanical complications | 12 months
  Complication rate with nail, cephalic screw, or distal screw
Parker mobility scale | 12 months
  Assessment of the patient's mobility capacity before and 12 months after hip surgery

CONTACTS AND LOCATIONS:
Overall Officials: Carlos De la Pinta Zazo, Principal Investigator — Elda University Hospital
Locations (1):
- Elda University Hospital, Elda, Valencia, Spain